CLINICAL TRIAL: NCT03340025
Title: Single-Use Negative Pressure Wound Therapy for Free Flap Donor Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Benjamin Greene, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300000596
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Surgical Wound
Keywords: negative pressure wound therapy; split thickness skin graft
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- negative pressure wound therapy (Experimental): PICO Single Use Negative Pressure Wound Therapy System
  Interventions: Device: PICO Single Use Negative Pressure Wound Therapy System
- conventional dressing (Placebo Comparator): traditional surgical wound dressing of xeroform gauze and padding
  Interventions: Device: xeroform gauze

INTERVENTIONS:
Device: PICO Single Use Negative Pressure Wound Therapy System — Class II negative pressure wound therapy powered suction pump
  Arms: negative pressure wound therapy
Device: xeroform gauze — traditional surgical dressing of xeroform gauze and padding
  Arms: conventional dressing

SUMMARY:
Various management options for free flap donor sites that require split thickness skin grafting exist. None has proven superior from both a patient care and a cost standpoint. Major complications occurring at these surgical sites include wound breakdown, tendon exposure, and loss of function. We seek to investigate the use of the PICO single-use negative pressure wound therapy device in these surgical sites and determine if it can yield superior results to simpler methods.

DETAILED DESCRIPTION:
Many studies have addressed the use of negative pressure wound therapy (NPWT) in free flap donor sites with mixed results. It is well established that NPWT is safe and causes no harm, and no delay in healing. A previous study performed at UAB showed that NPWT in complex Head & Neck Surgery reconstruction is safe, including free flap donor sites. There have been studies that state the rate of tendon exposure is lower with NPWT in free flap donor sites, and studies that conclude there is no difference in complication rates. Current clinical practice is varied, often within a single institution.

While no studies of NPWT in free flap donor sites have noted inferior results with its use, a primary reason cited for not using it is cost. Traditional NPWT using canister-based vacuum devices adds significant cost. The PICO single-use NPWT device (Smith & Nephew) is a relatively inexpensive, low-profile dressing that does not require attachment to an external canister. It is battery-powered and disposable. Empiric use on our patients undergoing split-thickness skin-grafting to free flap donor sites shows good results with minimal intra-operative effort compared to traditional bandaging. We would like to prospectively investigate the use of this low-cost NPWT device and compare it directly to the traditional post-op dressing method.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* participants are able to consent for themselves
* undergoing reconstructive surgery requiring split-thickness skin graft coverage of a free flap donor site (i.e., radial forearm free flap or fibula free flap)

Exclusion Criteria:

* < 18 years of age
* participants are unable to consent for themselves
* undergoing reconstructive surgery that does not require split-thickness skin graft coverage of a free flap donor site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Greene, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Negative Pressure Wound Therapy | Conventional Dressing
Started | 11 | 9
Completed | 9 | 7
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Pressure Wound Therapy | Conventional Dressing | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression of Wound Healing
Description: Comparison of photographs of all participants' wounds taken at post-operative Day 5, post-operative Day 14-21, and post-operative Day 30. Percentage skin graft take will be evaluated on Day 30 by blinded, independent raters. A 10x10 grid was digitally overlain on each image. The de-identified images were randomized and given to two independent raters. The raters used three criteria to assess each graft. Overall graft appearance was graded on a 1-5 scale, percent of graft take was estimated, and the presence of exposed tendon was noted for each timepoint.
Time Frame: Baseline through 30 days
Measure: Mean (Full Range); unit: percentage of skin graft take
Arm/Group | Negative Pressure Wound Therapy | Conventional Dressing
Number analyzed (Participants) | 9 | 7
percentage of skin graft take | 69.9 [50 to 90] | 75.6 [55 to 95]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Negative Pressure Wound Therapy | Conventional Dressing
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

LIMITATIONS AND CAVEATS:
The patient population is small. Our statistics indicate that assuming an 80% graft take, the number of patients needed for an appropriately powered study (80%) would be 44 patients in each group, while our study recruited only 9 and 11 patients to each group. This study is limited by missing data. Our study also takes place at a single center and, therefore, surgeon technique must be taken into account as this may have affected the outcomes of our data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT03340025/Prot_SAP_000.pdf